CLINICAL TRIAL: NCT02754947
Title: Etiology of Post-anesthetic and Post-sedation Events on the Inpatient Ward: Data From a Rapid Response Team at a Tertiary Care Children's Hospital
Brief Title: Need for the Assessment and Consultation Team (ACT) Following Anesthetic Care
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB14-00946
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Respiratory Diseases; Neurologic Diseases
Keywords: Assessment and Consultation Team (ACT); Rapid Response Team (RRT); Perioperative complications; Respiratory insufficiency; ASA status
MeSH Terms: conditions — Cardiovascular Diseases; Respiratory Tract Diseases; Nervous System Diseases; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study was to identify the etiology of events and demographics of patients that experience complications requiring activation of the Rapid Response Team (RRT) during the first 24 h following anesthetic care.

ELIGIBILITY:
Inclusion Criteria:

* Any study subject that experienced an ACT following anesthetic administration during care at any Nationwide Children's Hospital facility.

Exclusion Criteria:

* Any study subject that has not experienced an ACT following anesthetic administration during care at any Nationwide Children's Hospital facility.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any study subject that experienced an ACT following anesthetic administration during care at any Nationwide Children's Hospital facility reviewed from an existing Department of Anesthesiology & Pain Medicine database.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Identifying post-operative criteria for activation of Rapid Response Teams (RRTs) in caring for the pediatric population using Pediatric Early Warning Scores (PEWS) | 24 hours post-operatively
  To retrospectively identify the etiologies associated with a need to engage Rapid Response Teams (RRTs) to promote frequent assessments and early interventions among clinically deteriorating hospitalized pediatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: N'Diris Barry, BS, RN, MSN, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No